CLINICAL TRIAL: NCT07331350
Title: Effects of an Exercise Balance Program on Fall Prevention in Individuals With Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Exercise Balance Program for Fall Prevention in Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-17/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Accidental Falls; Balance Impairment; Physiotherapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly assigned to either an intervention group or a control group and will follow their respective exercise programs in parallel over the 5-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago-Based Balance Program With Additional Balance and Mobility Tasks (Experimental): Participants assigned to this arm will follow an Otago-based exercise program supplemented with additional balance and mobility tasks.
  Interventions: Other: Otago-Based Balance Program With Additional Balance and Mobility Tasks
- Otago Exercise Program (Active Comparator): Participants assigned to this arm will follow the Otago Exercise Program alone
  Interventions: Other: Otago Exercise Program only

INTERVENTIONS:
Other: Otago-Based Balance Program With Additional Balance and Mobility Tasks — Participants assigned to the intervention group followed a 5-week exercise-based balance program consisting of one supervised session per week combined with home-based exercises performed three times per week. The program was based on the Otago Exercise Program and was supplemented during supervised sessions with progressively challenging balance, mobility, and visuomotor tasks incorporating cognitive demands. Exercises included multidirectional stepping, lateral weight shifting, sit-to-stand movements, sideways walking, and heel-to-toe standing, with progression achieved through increased task complexity, speed, and duration. Additional task-oriented activities required participants to respond to verbal cues using colored floor markers to perform specific foot placements and postural tasks, with weekly variation in task-color associations to enhance cognitive engagement. A final multidirectional stepping task emphasized rapid changes in direction and movement speed, aiming to improve
  Arms: Otago-Based Balance Program With Additional Balance and Mobility Tasks
Other: Otago Exercise Program only — Participants assigned to the control group followed the Otago Exercise Program alone for a total duration of 5 weeks. The program consisted of standardized balance and lower-limb strengthening exercises designed for fall prevention and was performed exclusively as a home-based program three times per week. Exercises included multidirectional stepping, lateral weight shifting, sit-to-stand movements, sideways walking, and heel-to-toe standing, with progression achieved through adjustments in repetitions and sets. No supervised exercise sessions or additional balance, mobility, or cognitive tasks were provided to the control group during the intervention period.
  Arms: Otago Exercise Program

SUMMARY:
Falls are a major concern for individuals with Multiple Sclerosis (MS), negatively affecting balance, mobility, independence, and quality of life, while increasing the risk of injury. This randomized controlled trial aims to investigate the effects of a 5-week exercise-based balance program on fall-related outcomes in individuals with MS. Thirty participants with MS will be randomly allocated to either an intervention group or a control group. The intervention group will follow an Otago-based exercise program supplemented with additional balance and mobility tasks, while the control group will follow the Otago Exercise Program alone. Participants in both groups will perform home-based exercises three times per week. Outcomes will be assessed before and after the intervention period using the FICSIT-4 for balance, the Timed Up and Go test for mobility, the Falls Efficacy Scale-International (FES-I) for fear of falling, and the 12-item Multiple Sclerosis Walking Scale (MSWS-12) for walking limitations.

DETAILED DESCRIPTION:
Falls are a common and clinically significant problem in individuals with Multiple Sclerosis (MS), primarily associated with impairments in balance, mobility, muscle strength, and neuromuscular coordination. Exercise-based interventions focusing on balance and functional mobility constitute a core component of fall-prevention strategies; however, the optimal structure and intensity of such programs for individuals with MS remain under investigation.

This randomized controlled trial aims to investigate the effects of a 5-week exercise-based balance program on fall-related outcomes in individuals with MS. A total of 30 adults with a confirmed diagnosis of MS will be randomly allocated to either an intervention group or a control group using a parallel-group design.

Both groups will participate in a 5-week exercise program that includes home-based exercise performed three times per week. The control group will follow the Otago Exercise Program alone, a standardized and widely used balance and lower-limb strengthening program for fall prevention. The intervention group, in addition to performing the home-based Otago Exercise Program, will participate in one supervised exercise session per week. During these supervised sessions, the Otago-based program will be supplemented with additional balance and mobility tasks of progressively increasing difficulty, designed to challenge static and dynamic postural control, enhance neuromuscular coordination, and promote functional movement adaptability.

Outcome assessments will be conducted at baseline and immediately after completion of the intervention period. Balance will be assessed using the Four-Stage Balance Test (FICSIT-4), functional mobility will be evaluated with the Timed Up and Go test, fear of falling will be measured using the Falls Efficacy Scale-International (FES-I), and perceived walking limitations will be assessed using the 12-item Multiple Sclerosis Walking Scale (MSWS-12).

It is expected that participants in both groups will demonstrate improvements in balance and functional mobility following the intervention period, reflecting the effects of structured balance and strengthening exercises. It is further hypothesized that participants in the intervention group will exhibit greater improvements in balance performance and functional mobility compared with those in the control group, due to the addition of supervised balance and mobility tasks with increased task complexity. Reductions in fear of falling and perceived walking limitations are also anticipated, although these changes may be less pronounced than improvements observed in performance-based outcome measures.

The findings of this study are expected to contribute to a better understanding of exercise-based fall-prevention strategies for individuals with MS and to inform the design of targeted rehabilitation programs aimed at improving balance and mobility in this population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis.
* Ability to ambulate with or without an assistive device.
* Ability to understand and follow exercise instructions.
* Written informed consent prior to participation.

Exclusion Criteria:

* Presence of other neurological, musculoskeletal, or medical conditions that could significantly affect balance or mobility.
* Acute relapse of Multiple Sclerosis at the time of enrollment.
* Participation in another structured balance or fall-prevention program during the study period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Balance Performance (FICSIT-4) | Baseline and immediately after completion of the 5-week intervention
  Static balance will be assessed using the FICSIT-4 (Four-Stage Balance Test). Participants will attempt to maintain four progressively challenging standing positions (feet together, semi-tandem, tandem, and single-leg stance) for up to 10 seconds each, with eyes open and without an assistive device. The outcome will be recorded as the highest stage successfully held for 10 seconds (range: 0-4), with higher values indicating better balance performance.
Functional Mobility (Timed Up and Go Test) | Baseline and immediately after completion of the 5-week intervention
  Functional mobility will be assessed using the Timed Up and Go (TUG) test. Participants will be instructed to stand up from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down at a comfortable and safe pace. The time required to complete the task will be recorded in seconds. Shorter completion times indicate better functional mobility.
Fear of Falling (Falls Efficacy Scale-International) | Baseline and immediately after completion of the 5-week intervention
  Fear of falling will be assessed using the Falls Efficacy Scale-International (FES-I), a validated self-reported questionnaire consisting of 16 items that assess concern about falling during a range of daily activities. Each item is scored on a 4-point Likert scale, with total scores ranging from 16 to 64. Higher scores indicate greater concern about falling.
Walking Limitations (12-item Multiple Sclerosis Walking Scale) | Baseline and immediately after completion of the 5-week intervention
  Perceived walking limitations will be assessed using the 12-item Multiple Sclerosis Walking Scale (MSWS-12), a disease-specific, self-reported questionnaire that evaluates the impact of multiple sclerosis on walking ability. Items are scored on a Likert scale and transformed to a total score ranging from 0 to 100, with higher scores indicating greater walking impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Lytras, PhD, Principal Investigator — International Hellenic University
Locations (1):
- International Hellenic University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No